CLINICAL TRIAL: NCT03740945
Title: Effect of Intravaginal Prasterone (DHEA) on Moderate to Severe Symptoms of Vulvovaginal Atrophy Due to Menopause, in Women Under Treatment With an Aromatase Inhibitor for Breast Cancer - (Placebo-Controlled, Double Blind and Randomized Phase III Study)
Brief Title: Effect of Intravaginal Prasterone on Symptoms of VVA in Women Under Treatment With an Aromatase Inhibitor for Breast Cancer
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Business decision to not perform this study.
Sponsor: EndoCeutics Inc. (Industry)
Collaborators: AMAG Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ERC-260
Record Dates: First submitted 2018-11-07; First posted 2018-11-14 (Actual); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: Vaginal Atrophy in Breast Cancer Patients
Keywords: Vulvovaginal atrophy (VVA); Vaginal atrophy; Atrophic vaginitis; Prasterone; DHEA; Intrarosa; Breast cancer; Aromatase inhibitor
MeSH Terms: conditions — Atrophic Vaginitis; Breast Neoplasms | interventions — Dehydroepiandrosterone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo vaginal ovule daily for 12 weeks
  Interventions: Drug: Placebo
- Prasterone (Experimental): Prasterone (DHEA) vaginal ovule daily for 12 weeks
  Interventions: Drug: Prasterone (DHEA)

INTERVENTIONS:
Drug: Placebo — Daily administration of one placebo vaginal ovule at bedtime
  Arms: Placebo
Drug: Prasterone (DHEA) — Daily administration of one prasterone vaginal ovule at bedtime
  Other Names: Intrarosa
  Arms: Prasterone

SUMMARY:
The purpose of this study is to confirm the efficacy of intravaginal prasterone (DHEA) on moderate to severe (MS) and most bothersome symptoms (MBS) of vulvovaginal atrophy (VVA) due to natural, surgical or treatment-induced menopause, in women with breast cancer who are under treatment with an aromatase inhibitor.

ELIGIBILITY:
Inclusion Criteria:

Main criteria:

1. Natural, surgically- or treatment-induced postmenopausal women (non hysterectomized or hysterectomized) with breast cancer (stage 1 or 2) who is currently under treatment with an aromatase inhibitor and will remain on that treatment for the duration of the study.
2. Women between 30 and 80 years of age
3. Women having ≤5% of superficial cells on vaginal smear at baseline
4. Women having a vaginal pH above 5 at baseline
5. Women who have self-identified moderate or severe symptom(s) of vaginal atrophy

Exclusion Criteria:

Main criteria:

1. Clinically significant metabolic or endocrine disease (including diabetes mellitus) not controlled by medication
2. The administration of any investigational drug within 30 days of screening visit

Ages: 30 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-11-06 (Actual); Primary Completion 2019-12-05 (Actual); Study Completion 2019-12-05 (Actual)

PRIMARY OUTCOMES:
Change from Baseline to Week 12 in the Percentage of Superficial Cells | 12 weeks
Change from Baseline to Week 12 in the Percentage of Parabasal Cells | 12 weeks
Change from Baseline to Week 12 in Vaginal pH | 12 weeks
Change from Baseline to Week 12 in Moderate/Severe VVA symptom being Most Bothersome (MBS) | 12 weeks

SECONDARY OUTCOMES:
Change from Baseline to Week 12 in Moderate/Severe VVA symptom (not most bothersome) | 12 weeks
Change from Baseline to Week 12 on arousal/lubrication domain of Female Sexual Function Index (FSFI) questionnaire | 12 weeks
  Individual domain score will be obtained by adding the scores of the individual questions that comprise the domain and multiplying the sum by the domain factor.
Change from Baseline to Week 12 on subjective arousal domain of FSFI | 12 weeks
  Individual domain score will be obtained by adding the scores of the individual questions that comprise the domain and multiplying the sum by the domain factor.
Change from Baseline to Week 12 on desire domain of FSFI | 12 weeks
  Individual domain score will be obtained by adding the scores of the individual questions that comprise the domain and multiplying the sum by the domain factor.
Change from Baseline to Week 12 on satisfaction domain of FSFI | 12 weeks
  Individual domain score will be obtained by adding the scores of the individual questions that comprise the domain and multiplying the sum by the domain factor.
Change from Baseline to Week 12 on orgasm domain of FSFI | 12 weeks
  Individual domain score will be obtained by adding the scores of the individual questions that comprise the domain and multiplying the sum by the domain factor.
Change From Baseline to Week 12 in Severity of Vaginal Atrophy as Evaluated From Vaginal Secretions | 12 weeks
  Vaginal parameter evaluated at gynecological examination by the physician/gynecologist will be graded as corresponding to none, mild, moderate, or severe atrophy.
Change From Baseline to Week 12 in Severity of Vaginal Atrophy as Evaluated From Vaginal Epithelial Surface Thickness | 12 weeks
  Vaginal parameter evaluated at gynecological examination by the physician/gynecologist will be graded as corresponding to none, mild, moderate, or severe atrophy.
Change From Baseline to Week 12 in Severity of Vaginal Atrophy as Evaluated From Vaginal Epithelial Integrity | 12 weeks
  Vaginal parameter evaluated at gynecological examination by the physician/gynecologist will be graded as corresponding to none, mild, moderate, or severe atrophy.
Change From Baseline to Week 12 in Severity of Vaginal Atrophy as Evaluated From Vaginal Color | 12 weeks
  Vaginal parameter evaluated at gynecological examination by the physician/gynecologist will be graded as corresponding to none, mild, moderate, or severe atrophy.

CONTACTS AND LOCATIONS:
Overall Officials: Claude Labrie, M.D., Ph.D., Study Chair — Endoceutics, Inc., Quebec, Canada; David F Archer, M.D., Principal Investigator — Jones Institute, Norfolk VA 23507; Sheryl Kingsberg, Ph.D., Principal Investigator — MacDonald Women's Hospital, Cleveland, OH 44106 USA

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ke Y, Labrie F, Gonthier R, Simard JN, Bergeron D, Martel C, Vaillancourt M, Montesino M, Lavoie L, Archer DF, Balser J, Moyneur E; other participating Members of the Prasterone Clinical Research Group. Serum levels of sex steroids and metabolites following 12 weeks of intravaginal 0.50% DHEA administration. J Steroid Biochem Mol Biol. 2015 Nov;154:186-96. doi: 10.1016/j.jsbmb.2015.08.016. Epub 2015 Aug 17. PMID 26291918
- [Result] Labrie F, Derogatis L, Archer DF, Koltun W, Vachon A, Young D, Frenette L, Portman D, Montesino M, Cote I, Parent J, Lavoie L, Beauregard A, Martel C, Vaillancourt M, Balser J, Moyneur E; Members of the VVA Prasterone Research Group. Effect of Intravaginal Prasterone on Sexual Dysfunction in Postmenopausal Women with Vulvovaginal Atrophy. J Sex Med. 2015 Dec;12(12):2401-12. doi: 10.1111/jsm.13045. Epub 2015 Nov 23. PMID 26597311
- [Result] Labrie F, Montesino M, Archer DF, Lavoie L, Beauregard A, Cote I, Martel C, Vaillancourt M, Balser J, Moyneur E; other participating Members of the Prasterone Clinical Research Group. Influence of treatment of vulvovaginal atrophy with intravaginal prasterone on the male partner. Climacteric. 2015;18(6):817-25. doi: 10.3109/13697137.2015.1077508. Epub 2015 Oct 30. PMID 26517756
- [Result] Labrie F, Archer DF, Koltun W, Vachon A, Young D, Frenette L, Portman D, Montesino M, Cote I, Parent J, Lavoie L, Beauregard A, Martel C, Vaillancourt M, Balser J, Moyneur E; VVA Prasterone Research Group. Efficacy of intravaginal dehydroepiandrosterone (DHEA) on moderate to severe dyspareunia and vaginal dryness, symptoms of vulvovaginal atrophy, and of the genitourinary syndrome of menopause. Menopause. 2016 Mar;23(3):243-56. doi: 10.1097/GME.0000000000000571. PMID 26731686
- [Result] Martel C, Labrie F, Archer DF, Ke Y, Gonthier R, Simard JN, Lavoie L, Vaillancourt M, Montesino M, Balser J, Moyneur E; other participating members of the Prasterone Clinical Research Group. Serum steroid concentrations remain within normal postmenopausal values in women receiving daily 6.5mg intravaginal prasterone for 12 weeks. J Steroid Biochem Mol Biol. 2016 May;159:142-53. doi: 10.1016/j.jsbmb.2016.03.016. Epub 2016 Mar 10. PMID 26972555
- [Result] Montesino M, Labrie F, Archer DF, Zerhouni J, Cote I, Lavoie L, Beauregard A, Martel C, Vaillancourt M, Moyneur E, Balser J. Evaluation of the acceptability of intravaginal prasterone ovule administration using an applicator. Gynecol Endocrinol. 2016;32(3):240-5. doi: 10.3109/09513590.2015.1110140. Epub 2016 Jan 6. PMID 26634942
- [Result] Archer DF, Labrie F, Bouchard C, Portman DJ, Koltun W, Cusan L, Labrie C, Cote I, Lavoie L, Martel C, Balser J; VVA Prasterone Group. Treatment of pain at sexual activity (dyspareunia) with intravaginal dehydroepiandrosterone (prasterone). Menopause. 2015 Sep;22(9):950-63. doi: 10.1097/GME.0000000000000428. PMID 25734980
- [Result] Labrie F, Archer DF, Martel C, Vaillancourt M, Montesino M. Combined data of intravaginal prasterone against vulvovaginal atrophy of menopause. Menopause. 2017 Nov;24(11):1246-1256. doi: 10.1097/GME.0000000000000910. PMID 28640161